CLINICAL TRIAL: NCT00420303
Title: A Multicentre, Double-Blind, Placebo-Controlled, Randomized Study of Etanercept in the Treatment of Adults Patients With Refractory Heel Enthesitis in Spondylarthropathy
Brief Title: Study Evaluating Etanercept for the Treatment of Refractory Heel Enthesitis in Spondylarthropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A3-404
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Results first posted 2009-11-10 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Spondylarthropathies, Enthesitis
Keywords: Refractory Heel Enthesitis in Spondylarthropathy; Spondylarthropathy; Refractory Heel Enthesitis
MeSH Terms: conditions — Spondylarthropathies | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: Etanercept
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Etanercept — 50 mg injection once weekly
  Arms: A
Other: Placebo — placebo
  Arms: B

SUMMARY:
To assess the efficacy and safety of Etanercept in patients with spondylarthropathy and refractory heel enthesitis.

ELIGIBILITY:
Inclusion criteria

* Spondylarthropathy
* Heel enthesitis refractory to standard treatment
* Between 18 and 70 years of age
* The patient global assessment of the disease activity (measured by a 100 mm VAS) must be >40 in the last 48 hours

Exclusion criteria

* Use of > 1 local steroid injection within 2 weeks of screening
* Prior exposure to any TNF-inhibitor, including etanercept
* Dose of NSAIDs changed within two weeks of study drug evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com
Locations (15):
- France (12):
  - Arles
  - Avignon
  - Bordeaux
  - Grenoble
  - Montpellier
  - Nice
  - Orléans
  - Paris (Bichat)
  - Paris (cochin)
  - Paris (Pitie Salpetriere)
  - Strasbourg
  - Toulouse
- Germany (2):
  - Berlin
  - Herne
- Maastricht, Netherlands

REFERENCES:
- [Derived] Dougados M, Combe B, Braun J, Landewe R, Sibilia J, Cantagrel A, Feydy A, van der Heijde D, Leblanc V, Logeart I. A randomised, multicentre, double-blind, placebo-controlled trial of etanercept in adults with refractory heel enthesitis in spondyloarthritis: the HEEL trial. Ann Rheum Dis. 2010 Aug;69(8):1430-5. doi: 10.1136/ard.2009.121533. Epub 2010 May 28. PMID 20511606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from February 2007 to June 2008.
Pre-assignment Details: Patients were screened up to 6 weeks.
Groups:
- Etanercept: 50mg subcutaneously once weekly
- Placebo: Subcutaneously once weekly
Period: Overall Study
Arm/Group | Etanercept | Placebo
Started | 12 | 12
Completed | 11 | 8
Not Completed | 1 | 4
Not completed — Serious Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 34.5 (12.4) | 40.0 (10.4) | 37.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for Patient Global Assessment of Disease Activity (PGA) Between Randomization and Week 12
Description: PGA was measured using a 100mm Visual Analog Scale (VAS) ranging from 0=very good to 100=very bad. The normalized net incremental area under the curve of the PGA is the area between the baseline and the PGA curve as a function of time (week 2, 4, 8, 12). AUC was computed using the linear trapezoidal method. All the areas above the baseline and under the curve are positive and all the area below the baseline and above the curve are negative. The net incremental AUC is the sum of these areas. This result is then divided by the study duration of the patients. (negative value = improvement).
Time Frame: 12 weeks
Population: All randomized patients who received at least 1 dose of test article. Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 12 | 12
mm | -28.54 (18.01) | -11.07 (18.01)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Comparison of adjusted means; Test type: Superiority or Other; p = 0.029, ANCOVA; Treatment groups as fixed factors, baseline value as covariate; Mean Difference (Final Values) = -17.47, 95% CI [-32.93 to -2.01]

2. Secondary Outcome: Number of Patients Achieving a 50% Response on the Patient Global Assessment of Disease Activity
Description: A response is defined as at least a 50% improvement (decrease) from baseline in the patient global assessment of disease activity. The patient global assessment of disease activity was measured using a 100mm Visual Analog Scale (VAS) ranging from 0=very good to 100=very bad.
Time Frame: 12 weeks
Population: All randomized patients who received at least 1 dose of test article.
Measure: Number; unit: patients
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 12 | 12
patients | 8 | 2
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Test type: Superiority or Other; p = 0.02, Generalized estimating equations (GEE); Logit link, a binomial distribution and an auto-regressive correlation structure with treatment groups, visits and their interaction as fixed factors; Odds Ratio (OR) = 10.0, 95% CI [1.44 to 69.26]

3. Primary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity Score at Week 12
Description: The patient global assessment of disease activity was measured using a 100mm Visual Analog Scale (VAS) ranging from 0=very good to 100=very bad. Change=12 week score minus baseline score. A negative score indicates an improvement in disease activity and a positive score indicates worsening.
Time Frame: Baseline and 12 weeks
Population: All randomized patients who received at least 1 dose of test article.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 12 | 12
units on scale | -37.59 (22.04) | -11.58 (22.04)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA; Treatment groups, visits and their interaction as fixed factors, baseline value as a covariate and patients as a random factor

ADVERSE EVENTS:
Arm/Group | Etanercept | Placebo
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=12) | Placebo (N=12)
Cellulitis (Infections and infestations) | 1 | 0
Pharyngolaryngeal pain (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=12) | Placebo (N=12)
Chest pain (Cardiac disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 0
Injection site hypersensitivity (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1
Tracheitis (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Transaminases increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.